CLINICAL TRIAL: NCT05283135
Title: Decreasing Resident Memory T Cells While Increasing Clinical Durability: Higher Induction Doses of Risankizumab for Moderate-to-severe Plaque Psoriasis
Brief Title: High Dose Risankizumab for Psoriasis
Acronym: KNOCKOUT
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Oregon Medical Research Center (Other)
Collaborators: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: B20-433
Record Dates: First submitted 2022-02-03; First posted 2022-03-16 (Actual); Results first posted 2025-10-24 (Actual); Last update posted 2025-10-24 (Actual); Status verified 2025-10

CONDITIONS: Psoriasis
Keywords: Psoriasis; Risankizumab; Plaque; Skyrizi
MeSH Terms: conditions — Psoriasis; Plaque, Amyloid | interventions — risankizumab

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- risankizumab subcutaneous injection 600 mg (4x dosing) at Weeks 0, 4, and 16 (Experimental)
  Interventions: Drug: risankizumab
- risankizumab subcutaneous injection 300 mg (2x dosing) at Weeks 0, 4, and 16 (Experimental)
  Interventions: Drug: risankizumab

INTERVENTIONS:
Drug: risankizumab — Risankizumab (Skyrizi) is an anti-IL-23 antibody being investigated for the treatment of multiple inflammatory diseases, including psoriasis, Crohn's disease, ulcerative colitis, and psoriatic arthritis.
  Other Names: Skyrizi

SUMMARY:
This pilot study explores higher than standard doses of risankizumab for plaque psoriasis, to see effects on resident memory T cells and skin clearance.

DETAILED DESCRIPTION:
This is a pilot study that explores whether higher initial doses of risankizumab (300 mg and 600 mg, 2 times and 4 times the standard initial doses for plaque psoriasis) can more effectively target resident memory T cells, a type of immune cell within psoriatic lesions, and whether this results in higher levels of completely clear skin and for longer periods of time following withdrawal of drug. It is believed that resident memory T cells in psoriatic skin contribute to the persistence of psoriasis. It is believed that if the study drug can more effectively eliminate these cells, better clearance of psoriasis may be achieved (when compared to standard initial doses of study drug).

ELIGIBILITY:
Inclusion Criteria:

* Subject has provided written consent
* Subject has the ability to comply with all study visits and procedures
* Subject is at least 18 years of age
* Subject has chronic stable plaque psoriasis for at least 6 months and with a severity of BSA greater than or equal to 10 and PASI greater than or equal to 12
* Female subjects of child-bearing potential must have a negative urine test at screening and baseline. Female subjects must be either postmenopausal, or permanently surgically sterile, or for women of child-bearing potential practicing at least one form of birth control

Exclusion Criteria:

* Breastfeeding or pregnant women, or women who plan to become pregnant during study period
* Participation in any other clinical trial
* Active infection with HIV, hepatitis B virus, or hepatitis C virus
* Active infection with tuberculosis or untreated latent tuberculosis
* History of known active cancer, other than non-melanoma skin cancer or cervical carcinoma in situ, in the past 3 years
* History of drug or alcohol abuse in the past 6 months, as per investigator's assessment
* History of suicidal ideation or attempts in the past 6 months
* Presence of any concurrent illness, which in the opinion of the investigator, would place the patient at unnecessary safety risk during the trial or interfere with completion of the trial
* Treatment with topical medications for psoriasis in the past 2 weeks
* Treatment with oral medications for psoriasis in the past 4 weeks
* Phototherapy for psoriasis in the past 4 weeks
* Any prior treatment with Risankizumab
* Treatment with biologic medications for psoriasis (other than Risankizumab) in the past 4 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2022-03-01 (Actual); Primary Completion 2023-08-07 (Actual); Study Completion 2024-07-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin D Ehst, MD, PhD, Principal Investigator — Oregon Medical Research Center
Locations (1):
- Oregon Medical Research Center, Portland, Oregon, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gordon KB, Strober B, Lebwohl M, Augustin M, Blauvelt A, Poulin Y, Papp KA, Sofen H, Puig L, Foley P, Ohtsuki M, Flack M, Geng Z, Gu Y, Valdes JM, Thompson EHZ, Bachelez H. Efficacy and safety of risankizumab in moderate-to-severe plaque psoriasis (UltIMMa-1 and UltIMMa-2): results from two double-blind, randomised, placebo-controlled and ustekinumab-controlled phase 3 trials. Lancet. 2018 Aug 25;392(10148):650-661. doi: 10.1016/S0140-6736(18)31713-6. Epub 2018 Aug 7. PMID 30097359
- [Background] Reich K, Gooderham M, Thaci D, Crowley JJ, Ryan C, Krueger JG, Tsai TF, Flack M, Gu Y, Williams DA, Thompson EHZ, Paul C. Risankizumab compared with adalimumab in patients with moderate-to-severe plaque psoriasis (IMMvent): a randomised, double-blind, active-comparator-controlled phase 3 trial. Lancet. 2019 Aug 17;394(10198):576-586. doi: 10.1016/S0140-6736(19)30952-3. Epub 2019 Jul 4. PMID 31280967
- [Background] Blauvelt A, Leonardi CL, Gooderham M, Papp KA, Philipp S, Wu JJ, Igarashi A, Flack M, Geng Z, Wu T, Camez A, Williams D, Langley RG. Efficacy and Safety of Continuous Risankizumab Therapy vs Treatment Withdrawal in Patients With Moderate to Severe Plaque Psoriasis: A Phase 3 Randomized Clinical Trial. JAMA Dermatol. 2020 Jun 1;156(6):649-658. doi: 10.1001/jamadermatol.2020.0723. PMID 32267471

RESULTS

PARTICIPANT FLOW:
Groups:
- 600 mg Dose Group: Received risankizumab subcutaneous injection 600 mg (4x dosing) at Weeks 0, 4, and 16 and then no further injections. Subjects were followed through week 100, the first 52 weeks in a double-blind manner, then the next 48 weeks in an unblinded extension period.
- 300 mg Dose Group: Received risankizumab subcutaneous injection 300 mg (2x dosing) at Weeks 0, 4, and 16 and then no further injections. Subjects were followed through week 100, the first 52 weeks in a double-blind manner, then the next 48 weeks in an unblinded extension period.
Period: Overall Study
Arm/Group | 600 mg Dose Group | 300 mg Dose Group
Started | 10 | 10
Completed Dosing (Week 16) | 9 | 9
Completed 52 Week Blinded Period | 8 | 8
Completed | 3 | 3
Not Completed | 7 | 7

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 600 mg Dose Group | 300 mg Dose Group | Total
Number analyzed (Participants) | 10 | 10 | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.9 (16.3) | 48.7 (13.0) | 46.8 (14.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 3 | 7
  Male | 6 | 7 | 13
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 3 | 3
  Not Hispanic or Latino | 10 | 7 | 17
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 1 | 2
  White | 8 | 8 | 16
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Psoriasis disease duration [Mean (Standard Deviation); unit: years] | 26.0 (18.1) | 16.9 (15.1) | 21.4 (16.9)
Weight [Mean (Standard Deviation); unit: kg] | 88.42 (20.7) | 86.7 (13.7) | 87.6 (17.1)
sPGA [Count of Participants; unit: Participants] — The static Physician's Global Assessment (sPGA) is a 5-point scale ranging from 0 to 4 (0=clear, 1=almost clear, 2=mild, 3=moderate, and 4=severe). Scores are assigned based on the Investigator's assessment of the average erythema, thickness and scale of all psoriasis plaques at a given timepoint, without consideration of prior timepoints (hence "static").
  Participants
    sPGA 3 (moderate) | 4 | 9 | 13
    sPGA 4 (severe) | 6 | 1 | 7

OUTCOME MEASURES:

1. Primary Outcome: CD8+ Trm1 Cells in Lesional Skin at Baseline and Week 52
Description: The number of lesional CD8+ Trm1 cells at baseline and Week 52 was calculated by longitudinal single-cell RNA-sequencing of full-thickness skin biopsy samples. Uniform Manifold Approximation Projection (UMAP) was used for T cell subtype visualization and CD8+ Trm1 cells were identified as IFNγ+/CD8+/CD69+ T cells.
Time Frame: 52 weeks
Population: Cell counts from all participants were analyzed together at baseline given the exploratory nature of this study, the small number of overall participants and the selection of trial participants on the basis of clinical parameters that assume a similar degree of memory cell infiltrate in lesional psoriasis plaques.
Measure: Mean (95% Confidence Interval); unit: number of cells
Groups:
- 600 mg Baseline; 600 mg Week 52; 300 mg Week 52: Lesional skin from those participants who received risankizumab subcutaneous injection 600 mg (4x dosing) at Weeks 0, 4, and 16 and then no further injections.
- 300 mg Baseline: Lesional skin from those participants who received risankizumab subcutaneous injection 300 mg (4x dosing) at Weeks 0, 4, and 16 and then no further injections.
Arm/Group | 600 mg Baseline | 300 mg Baseline | 600 mg Week 52 | 300 mg Week 52
Number analyzed (Participants) | 5 | 8 | 5 | 8
number of cells | 9.60 [-1.97 to 21.17] | 26.71 [7.00 to 46.43] | 1.60 [0.18 to 3.02] | 16.63 [0.15 to 33.10]

2. Primary Outcome: CD8+ Trm17 Cells in Lesional Skin at Baseline and Week 52
Description: The number of lesional CD8+ Trm17 cells at baseline and Week 52 was calculated by longitudinal single-cell RNA-sequencing of full-thickness skin biopsy samples. Uniform Manifold Approximation Projection (UMAP) was used for T cell subtype visualization and CD8+ Trm17 cells were identified as IFNγ+/CD8+/CD69+ T cells.
Time Frame: 52 weeks
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: number of cells
Arm/Group | 600 mg Baseline | 300 mg Baseline | 600 mg Week 52 | 300 mg Week 52
Number analyzed (Participants) | 5 | 8 | 5 | 8
number of cells | 19.67 [-28.52 to 67.86] | 22.88 [5.94 to 39.81] | 3.20 [-5.01 to 11.41] | 5.00 [-1.00 to 11.00]

3. Secondary Outcome: PASI 100 Results in Patients Receiving 4X Standard Induction Doses of Risankizumab vs. Those Receiving 2X Standard Induction Doses of Risankizumab.
Description: The percentage of patients with Psoriasis Area and Severity Index (PASI) 100 (complete clearance) at Weeks 28, 40, and 52 in patients receiving 4X standard induction doses of risankizumab vs. those receiving 2X standard induction doses of risankizumab.
Time Frame: Enrollment to Week 52
Population: 18 total subjects completed all 3 risankizumab injections and were considered evaluable in efficacy assessments
Measure: Count of Participants; unit: Participants
Arm/Group | 600 mg Dose Group | 300 mg Dose Group
Number analyzed (Participants) | 9 | 9
Participants
  PASI 100 at week 28 | 7 | 8
  PASI 100 at week 40 | 6 | 6
  PASI 100 at week 52 | 4 | 4

4. Secondary Outcome: Safety Events
Description: Safety events over 52 weeks in patients receiving 4X standard induction doses of risankizumab vs. those receiving 2X standard induction doses of risankizumab.
Time Frame: Enrollment to Week 52
Population: Treatment emergent adverse events
Measure: Number; unit: events
Arm/Group | 600 mg Dose Group | 300 mg Dose Group
Number analyzed (Participants) | 10 | 10
events
  TEAE | 11 | 11
  TEAE related to study treatment | 0 | 0
  Serious or severe TEAE | 0 | 1
  Serious TEAE related to study treatment | 0 | 0

ADVERSE EVENTS:
Time Frame: 100 weeks
Description: AEs were collected from the time of consent at all subject visits
Arm/Group | 600 mg Dose Group | 300 mg Dose Group
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10 | 1/10
Other Adverse Events (participants affected / at risk) | 7/10 | 9/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 600 mg Dose Group (N=10) | 300 mg Dose Group (N=10)
worsening right tibial fracture and meniscal tear (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) — seriousness based on hospitalization
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 600 mg Dose Group (N=10) | 300 mg Dose Group (N=10)
COVID-19 infection (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1)
Common cold (Respiratory, thoracic and mediastinal disorders) | 3 (4) | 1 (1)
Eczematous dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Hyperglycemia (Endocrine disorders) | 0 (0) | 1 (1)
Bleeding internal hemorrhoids (Gastrointestinal disorders) | 0 (0) | 1 (1)
Bursitis, left elbow (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Worsening psoriatic arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Neutrophilia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Osteoarthritis, right hip (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Worsening osteoarthritis, right hip (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Cellulitis, left lower extremity (Infections and infestations) | 1 (1) | 0 (0)
Hypercholesterolemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Transaminitis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Low back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Right tibial fracture and meniscal tear (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Left inguinal hernia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (2) | 0 (0)
Gastroenteritis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Worsening glaucoma (Eye disorders) | 1 (1) | 0 (0)
Upper respiratory infection (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 2 (3)
Cough (General disorders) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
Small sample size

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-02-22): https://cdn.clinicaltrials.gov/large-docs/35/NCT05283135/Prot_SAP_000.pdf